CLINICAL TRIAL: NCT02682966
Title: Direct Evaluation of Postoperative Myocardial Injury Using Coronary Computed Tomography Angiography After Non-Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Wilton A van Klei, Prof. dr., UMC Utrecht
Other Study IDs: DEPICT-NCS
Record Dates: First submitted 2016-02-03; First posted 2016-02-17 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Myocardial Injury
Keywords: troponin; coronary artery disease; pulmonary embolism; Computed Tomography Angiography; postoperative myocardial injury
MeSH Terms: conditions — Coronary Artery Disease; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PMI: Postoperative Myocardial injury, postoperative troponin levels ≥ 60 ng/L
  Interventions: Radiation: Coronary Computed Tomography Angiography
- Control: postoperative troponin levels < 60 ng/L
  Interventions: Radiation: Coronary Computed Tomography Angiography

INTERVENTIONS:
Radiation: Coronary Computed Tomography Angiography — Coronary Computed Tomography Angiography will be performed in all participants

SUMMARY:
This is a prospective study in patients who undergo routine postoperative troponin assessment after major (semi-)elective noncardiac surgery. Two groups are created based on postoperative troponin levels: Postoperative myocardial injury (PMI) group with troponin I levels ≥ 60 ng/L and a control group with troponin levels < 60ng/L. The primary aim of this study is to assess the association of PMI with pulmonary embolism. Additionally, the association between PMI and obstructive CAD will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years old
* Major noncardiac surgery, defined as non-cardiac surgical procedures requiring hospital admittance > 24 hours
* Semi-elective surgery, defined as surgery that that has been preceded by a preoperative evaluation.
* ≥ 1 troponin assessment in the first 3 postoperative days as a part of the routine 'postoperative troponin assessment' protocol.
* For patients who undergo surgery more than once, the first surgery will be included in the analysis. Reoperations will not be included.

Exclusion Criteria:

* Typical anginal complaints
* Acute ST-elevation myocardial infarction (STEMI) or new left bundle branch block (LBBB) on ECG
* Patients unable to fully comply to study needs (e.g. incompetent patients or patients unable to communicate in Dutch or English)
* Severe claustrophobia.
* Patients who have a life expectancy of less than three months.
* Patients who are too ill to undergo a CCTA or Ventilation/Perfusion (V/Q) scan.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 60 years or older that undergo major (semi-)elective noncardiac surgery are eligible for study participation. Major (semi)-elective noncardiac surgery is defined as all surgical procedures requiring ≥ 24 hours of hospital admittance that have been preceded by a preoperative evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Embolism | 1 week
  Pulmonary embolism (PE) on either Coronary Computed Tomography Angiography (CCTA) or Ventilation/Perfusion (V/Q) scan. PE on CCTA is defined as a sharply delineated pulmonary artery filling defect in at least two consecutive image sections of the CCTA, either located centrally within the vessel or with acute angles at its interface with the vessel wall. PE on V/Q scan is defined as at least one segmental or two subsegmental perfusion defects without corresponding abnormality on chest X-ray.

SECONDARY OUTCOMES:
Obstructive coronary artery disease | 1 week
  > 50% stenosis in one or more epicardial vessels on CCTA
Obstructive main stem or proximal left anterior descending (LAD) stenosis | 1 week
  Incidence of obstructive (>50%) main stem or proximal left anterior descending (LAD) stenosis
30-day MACE | 30 days
  Major adverse cardiovascular events within 30 postoperative days, which is defined as the composite of cardiovascular death, non-fatal myocardial infarction, non-fatal cardiac arrest, non-fatal ventricular fibrillation and ventricular arrhythmia with hemodynamic compromise.
30-day all-cause mortality | 30-day
major diagnostic changes | 1 week
  Major Diagnostic change, which is defined as a clinically relevant change in diagnosis after CCTA in comparison to the most likely diagnosis before CCTA. The diagnosis prior to CCTA is made by the cardiology consultant and is based on routine clinical
major therapeutic changes | 1 week
  Major Therapeutic change, which is defined as any change in in management of patients due to CCTA findings compared to the proposed treatment before CCTA
bleeding | 1 year after surgery
  bleeding within one year after surgery, which is based on TIMI criteria

CONTACTS AND LOCATIONS:
Overall Officials: Wilton A van Klei, MD, PhD, Principal Investigator — UMC Utrecht

IPD SHARING:
Plan to Share IPD: Undecided